CLINICAL TRIAL: NCT06991322
Title: Self-Expanding Coronary Sinus Reducer for Treatment of Symptomatic Coronary Microvascular Dysfunction (CMD) (SERRA-I Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VahatiCor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VHC-00002
Record Dates: First submitted 2025-05-19; First posted 2025-05-27 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Coronary Microvascular Dysfunction; Coronary Microvascular Disease
MeSH Terms: conditions — Microvascular Angina

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Other)
  Interventions: Device: A-FLUX Reducer System

INTERVENTIONS:
Device: A-FLUX Reducer System — The VahatiCor A-FLUX Reducer System is an implantable, self-expanding dense-cell nitinol coronary sinus flow restrictor device pre-loaded into the A-FLUX Delivery Catheter.

SUMMARY:
VahatiCor's Coronary Sinus Reducer (A-FLUX) has been designed to improve angina or angina-like symptoms in patients with CMD. SERRA-I is an early feasibility study that evaluates the safety and clinical performance of the A-FLUX Reducer in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years of age.
2. Left ventricular ejection fraction (LVEF) is greater than or equal to 25% within the 12 months before the index procedure.
3. Greater than or equal to 30 days of persistent symptomatic coronary microvascular dysfunction (angina pectoris, or equivalent symptoms) (classified as CCS Grade II-IV angina, or NYHA Class 2 or 3 equivalent non-anginal functional impairment) despite optimal medical therapy as determined by Investigator and confirmed by the Central Screening Committee.
4. CFR<2.5 measured with continuous thermodilution within 30 days of index procedure.
5. Sustained angina (or equivalent symptoms) reported for at least 2 weeks leading up to the index procedure, as reported via the ORBITA-app.
6. Willing and able to sign informed consent.
7. Willing to comply with the specified follow-up evaluations.
8. Mean right atrial pressure ≤15 mmHg.
9. The CS anatomy is suitable for implantation at the Investigator's discretion.

Exclusion Criteria:

1. Significant obstructive epicardial disease (greater than 50% diameter stenosis) that can be treated with PCI or CABG as determined by Investigator and confirmed by the Central Screening Committee.
2. Recent (less than 30 days before index procedure) troponin or CKMB positive acute coronary syndrome (NSTEMI or STEMI) with evidence of ischemia.
3. Extra-coronary contributory causes of angina - e.g., untreated hyperthyroidism, anemia (Hgb less than 9 g/dL), uncontrolled hypertension (systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than 100 mmHg despite medications), atrial fibrillation with a rapid ventricular response (consistently greater than 100 bpm despite medications) or other tachyarrhythmia, severe aortic stenosis, decompensated heart failure, hypertrophic cardiomyopathy with left ventricular outflow tract obstruction or asymmetric septal hypertrophy (concentric left ventricular hypertrophy is not an exclusion criterion).
4. NYHA class IV or decompensated HF or hospitalization due to HF during the 90 days before the index procedure.
5. Life-threatening rhythm disorders or any rhythm disorders that would require cardiac resynchronization therapy or lead placement in the coronary sinus.
6. Severe chronic obstructive pulmonary disease (COPD) as indicated by a forced expiratory volume in one second (FEV1) of less than 1.0L or need for home daytime oxygen or regular oral steroids.
7. Severe valvular heart disease (any valve).
8. Moderate (TAPSE<12) or severe RV dysfunction (TAPSE<8) by echocardiography.
9. A pacemaker electrode/lead is present in the coronary sinus.
10. Recent implantation of a new pacemaker or defibrillator leads with any electrode in the right atrium within 90 days of the index procedure.
11. Chronic severe renal failure (estimated eGFR less than 30 mL/min/1.73m2 or equivalent) or subjects on chronic dialysis.
12. Known allergy to titanium, nickel, platinum, tungsten or known inability to tolerate contrast medium.
13. Any clinical condition that might interfere with the trial protocol or the subject's ability to be compliant with the trial protocol (e.g., active alcohol or illicit substance use, cognitive decline).
14. Currently enrolled in another investigational device or drug trial that has not reached its primary endpoint or might clinically interfere with the current trial endpoints or procedures.
15. Pregnant or planning pregnancy within the next 12 months (females of reproductive potential must have a negative pregnancy test within 7 days of the procedure).
16. Part of a vulnerable population who, in the investigator's judgment, cannot give Informed Consent for reasons of incapacity, immaturity, adverse personal circumstances, or lack of autonomy.
17. Inability to tolerate dual antiplatelet therapy for 6 months if not on a chronic oral anticoagulant, or inability to tolerate a P2Y12 inhibitor for at least 6 months if on a chronic oral anticoagulant.
18. Comorbidities limiting life expectancy to less than one year.
19. Currently hospitalized for definite or suspected COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Procedural Success | Throughout the study, up to 12 months post-procedure
  Successful delivery and deployment of VahatiCor A-FLUX Reducer System
Safety: Rate of device- and procedure- related SAEs | 30-days post-procedure
  Rate of device- and procedure-related SAEs.

CONTACTS AND LOCATIONS:
Locations (2):
- University Medical Center Utrecht, Utrecht, Netherlands
- Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu, Warsaw, Poland